CLINICAL TRIAL: NCT06211439
Title: Clinical Study on Efficacy and Mechanism of HD-tACS in Patients With Prolonged Disorders of Consciousness
Brief Title: Transcranial Alternating Current Stimulation in Patients With Disorders of Consciousness
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: tACS in pDoC
Record Dates: First submitted 2024-01-08; First posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2023-05

CONDITIONS: Consciousness Disorders
Keywords: disorders of consciousness; Transcranial alternating current stimulation; tACS; EEG
MeSH Terms: conditions — Consciousness Disorders

STUDY DESIGN:
Intervention Model Description: Using a sham-controlled randomized double-blind design, 64 patients were randomly assigned to either a real or sham stimulation group. In the real stimulation group, stimulation of different frequencies (40Hz gamma, 4Hz theta) is applied to the left dorsolateral prefrontal cortex with a current intensity of 2mA for 20 minutes each day, continuously for 5 days. In the sham stimulation group, the tACS stimulation mode and frequency are the same as in the real stimulation group, but current is only applied during the first and last 30 seconds of the entire 20-minute stimulation period.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcranial electrical stimulation HD-tES (Active Comparator): real HD-tACS:anodal transcranial alternating current stimulation were delivered over the left DLPF cortex for patients in different frequencies (40Hz gamma, 4Hz theta) , with a current intensity of 2mA for 20 minutes per day.
  Interventions: Device: real transcranial alternating current stimulation
- sham Transcranial electrical stimulation HD-tES (Sham Comparator): sham HD-tACS: sham transcranial alternating current stimulation were delivered over the left DLPF cortex for patients in different frequencies (40Hz gamma, 4Hz theta) , with a current intensity of 2mA for 20 minutes per day.
  Interventions: Device: sham transcranial alternating current stimulation

INTERVENTIONS:
Device: real transcranial alternating current stimulation — The alternating current was non-invasively delivered using an M×N five-channel high-definition transcranial electrical current stimulator (Soterix Medical). A BrainCap (Brain Vision) embedded with high-definition plastic holders consisted of five 12-mm-diameter Ag/AgCl ring electrodes, filled with conductive gel. During real HD-tACS, the current was increased to 2 mA from the onset of stimulation and applied for 20 minutes.
  Arms: Transcranial electrical stimulation HD-tES
Device: sham transcranial alternating current stimulation — For the sham condition(sham HD-tACS), the same electrode placement was used as in the stimulation condition, but the current was only applied during the first and last 30 seconds of the entire 20-minute stimulation period.
  Arms: sham Transcranial electrical stimulation HD-tES

SUMMARY:
In recent years, many literatures have reported that tACS, as a non-invasive electrical brain stimulation technique, has been applied in depression, schizophrenia, dementia and other fields.

The goal of this study is to explore the clinical efficacy and mechanism of action of HD-tACS in patients with chronic disorders of consciousness.The main questions it aims to answer are:

1. Explore the neurophysiological effects of HD-tACS on patients with chronic disorders of consciousness under theta and gamma frequency stimulation, and observe its impact on behavioral changes and long-term prognosis;
2. Further investigate the awakening mechanism of consciousness disorders through HD-tACS stimulation using multimodal assessment;
3. Clarify the role of theta and gamma neural oscillations in consciousness disorders, providing new targets for the pathogenesis and treatment of Disorders of Consciousness .

DETAILED DESCRIPTION:
Background: tACS is a transcranial nerve regulation technique ,it has been applied in depression, schizophrenia, dementia and other fields. However, the exact mechanism of tACS has not been fully elucidated, and there are few reports about the effect of tACS stimulation on patients with consciousness disorder at home and abroad.

Objective: The study aimed to investigate the reactivity of electroencephalography (EEG) and the clinical response of patients with disorders of consciousness and explore the neuromodulatory effects of HD-tACS in patients with chronic disorders of consciousness.

Method: Based on inclusion and exclusion criteria, patients with disorders of consciousness are categorized into chronic coma, vegetative state (VS), and minimally conscious state (MCS) groups. General and clinical data of the patients are collected. Assessments using the CRS-R scale and resting-state EEG are conducted before and after the trial. The trial is designed as a randomized controlled experiment, divided into an HD-tACS real stimulation group and a sham stimulation group. In the real stimulation group, different frequencies (40Hz gamma, 4Hz theta) of stimulation are applied to the left dorsolateral prefrontal cortex, with a current intensity of 2mA for 20 minutes per day, continuously for 5 days. In the sham stimulation group, the tACS stimulation mode and frequency are consistent with the real stimulation group, but current is only passed during the first and last 30 seconds of the entire 20-minute stimulation period. EEG is collected for all patients before stimulation, on the first day of stimulation, and after the stimulation ends. Follow-ups include CRS-R scale and GOS-E scores after 3 months and GOS-E scores after 6 months.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients with consciousness disorders for more than 28 days following severe brain injury, assessed by the CRS-R scale to meet the criteria for VS or MCS; 2. Aged between 14 and 80 years; 3. Stable vital signs; 4. No neuromuscular function blockers and no sedation within the prior 24 hours;

Exclusion Criteria:

* 1. Locked-in syndrome; 2. Contraindications for EEG examination;HD-tACS stimulation. 3. Contraindications for MRI scanning, such as the presence of internal metallic implants; 4. Diseases and factors that may affect brain function assessment, such as metabolic disorders, poisoning, shock, etc.

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2022-12-05 (Actual); Primary Completion 2024-05-10 (Estimated); Study Completion 2024-10-31 (Estimated)

PRIMARY OUTCOMES:
the JFK Coma Recovery Scale-Revised (CRS-R) scale | at baseline (T0), immediately after the end of the treatment (T1), 5 days later (T2).Investigators observed the changes from baseline to the end of stimulation
  The primary outcome measure is the change in the CRS-R scale in patients with prolonged Disorders of Consciousness (pDoC) after 5 days of HD-tACS treatment.The CRS-R is a tool used to characterise the level of consciousness.The CRS-R is a tool used to characterize the level of consciousness and to monitor neurobehavioural recovery in DOC. The scale consists of 23 hierarchically arranged items that comprise six subscales addressing the auditory, visual, motor, oromotor/verbal, communication and arousal processes. The lowest item on each subscale represents reflexive activity whereas the highest item represents cognitively mediated behaviors

SECONDARY OUTCOMES:
EEG data ( electrophysiological parameters) | at baseline (T0), immediately after the end of the treatment (T1), 5 days later (T2)
  delta (1-4 Hz), theta (4-8 Hz), alpha (8-12 Hz) and beta (12-30 Hz).an increase of delta and theta activity usually reflects encephalopathy and/or structural lesions, interpreted as poor outcome predictor of DOC .The power of α and β is related to the chance of recovery.

OTHER OUTCOMES:
Glasgow Outcome Scale-Extended (GOS-E) | In the first and third months after the stimulus ends
  GOS-E is an extended version of the Glasgow Outcome Scale (GOS), which was developed to provide a more detailed assessment of patient functionality and quality of life after experiencing brain injury. It has eight categories:Dead, Vegetative State, Lower Severe Disability, Upper Severe Disability, Lower Moderate Disability, Upper ModerateDisability, Lower Good Recovery, and Upper Good Recovery.Percentage of patients with improved consciousness (GOS-E score improved by 1 point or more) three months after stimulation ended.

CONTACTS AND LOCATIONS:
Overall Officials: Benyan Luo, Prof, Dr, Principal Investigator — The First Affiliated Hospital, Zhejiang University
Locations (1):
- The First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No